CLINICAL TRIAL: NCT04424355
Title: Possibilities of Chest Magnetic Resonance Imaging (MRI) in Diagnostics of COVID-19. The Use of MRI to Assess Lung Damage in Patients With Coronavirus Infection
Brief Title: Magnetic Resonance Imaging to Detect Signs of Viral Pneumonia in Patients With Coronavirus Infection.
Status: Completed | Type: Observational
Sponsor: Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department (Other)
Responsible Party: Principal Investigator, Sergey Morozov, Chief Research Officer, Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department
Other Study IDs: 2020-2
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Coronavirus Infections; Pneumonia
Keywords: Computed tomography; Magnetic resonance imaging; Lung MRI
MeSH Terms: conditions — Coronavirus Infections; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with suspected pneumonia COVID-19: Chest MRI findings: bilateral, diffuse ground-glass opacity (GGO), consolidation, "crazy paving" pattern, pleuritis.
- Patients with suspected pneumonia with COVID -19: Chest CT findings: bilateral, diffuse ground-glass opacity (GGO), consolidation, "crazy paving" pattern, pleuritis.
  Interventions: Diagnostic Test: Chest MRI

INTERVENTIONS:
Diagnostic Test: Chest MRI — Patients referred by the primary care physician with suspected pneumonia
  Other Names: Chest CT scan
  Groups: Patients with suspected pneumonia with COVID -19

SUMMARY:
Since the onset of the COVID-19 pandemic, the importance of chest computed tomography (CT) in detecting signs of viral pneumonia has become clear from the literature. However, the increased patient flow creates an additional pressure on CT centers. We believe, the use of chest magnetic resonance imaging (MRI) can help to test patients for CОVID-19 when CT scan is not available. Lung MRI may be useful in routing a patient in a difficult epidemiological situation.

DETAILED DESCRIPTION:
Currently, with increased load of CT studies, alternative methods of viral pneumonia signs' visualization are required.

Investigators hypothesize that chest MRI could be a test for detecting pulmonary features of COVID-19. They consider using MRI to assess COVID-19 viral pneumonia. Absence of radiation exposure to patients is a clear advantage of MRI.

This is a prospective, observational cohort study assessing patients with suspected COVID-19. It's primary goal is to determine the ability of multiparametric MRI to detect lung abnormalities - ground-glass opacity (GGO), consolidation, "crazy paving" pattern, pleuritis - in comparison to CT scan. In this study each patient with suspected pneumonia will sequentially undergo both chest CT and MRI during his/her visit. Scan protocols will be identical for each patient. Each participants completed an online questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* A referral from the attending physician for a chest CT scan
* Suspected pneumonia
* Signed informed consent
* Over 18 years old

Exclusion Criteria:

* Pregnant or nursing women
* Presence of foreign implanted objects in the body at the scan level (including cardiac pacemakers, spine metalware)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with suspected viral COVID-19 pneumonia will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Number of zones of pulmonary parenchyma corresponding to viral pneumonia detected by chest MRI in comparison with CT scan | Upon completion, up to 1 year
  Expected number - more than two zones

CONTACTS AND LOCATIONS:
Locations (1):
- Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No